CLINICAL TRIAL: NCT05076305
Title: PelvEx 4: Advanced Pelvic Malignancy and the Role of the Multi-disciplinary Team Meeting - An International Assessment of MDT Decisions
Brief Title: PelvEx 4: Advanced Pelvic Malignancy and the Role of the Multi-disciplinary Team Meeting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St Vincent's University Hospital, Ireland (Other)
Collaborators: PelvEx collaborative (Unknown)
Responsible Party: Principal Investigator, Professor Des Winter, Consultant Gastrointestinal Surgeon, St Vincent's University Hospital, Ireland
Other Study IDs: STVINCENTS
Record Dates: First submitted 2021-04-19; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Multidisciplinary Communication; Locally Advanced Rectal Cancer; Recurrent Rectal Cancer; Multidisciplinary Team Meeting (MDT); Treatment Decisions
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No specific intervention; cases are retrospective and patients have already been treated. — To assess the geographic variation that exists in the management of locally advanced and recurrent rectal cancers.

SUMMARY:
The treatment of locally advanced and recurrent rectal cancers is highly individualized to each patient and their pattern of disease, and this decision is often made at the Multidisciplinary Team (MDT) meeting . The PelvEx collaborative was designed with the intent to provide greater international consensus on appropriate treatment decisions for this cohort. However, we propose that international variation exists in how certain patients will be evaluated, assessed and ultimately treated despite having the same disease. We plan to measure this variation in order to provide a greater understanding of the differences that exist.

DETAILED DESCRIPTION:
The PelvEx collaborative is an international research collaborative that was designed with the aim of collating data on patients undergoing pelvic exenteration from all corners of the globe. These extensive procedures, despite their associated morbidity, have revolutionised the approach to advanced pelvic malignancy and provide hope to patients whose cancers would have once been deemed inoperable. Despite the increasing frequency with which surgeons are performing these more radical resections (1), relatively few of these procedures are carried out when compared with more traditional surgical operations. Furthermore, this cohort of patients and the wide-ranging procedures which they undergo represent a heterogenous group. These factors combine to make it more difficult for academic surgeons to draw meaningful conclusions from their study, and further illustrate the need for prospective international collaboration in order to inform appropriate treatment strategies.

However, despite the great demand for international collaboration, it is vital that there is an appreciation of the variation in the approach to managing these complex cases between hospitals, countries and continents. While surgeons would like to believe that in any case where their local multi-disciplinary team meeting has made an informed treatment decision that it is the single most appropriate option, geographic variation in beliefs, attitudes, terminology and patient preferences may influence those decisions at an individual level. Nowhere is this more relevant than in the approach to advanced pelvic malignancy. One study analysing regional variation in the management of locally advanced and recurrent rectal cancer noted a significantly lower rate of pelvic exenteration in France when compared with Australia, despite intercountry blinding of radiological findings (2). These differences are influenced by a host of psychosocial factors that are as yet to be fully elucidated.

The goal of the present analysis is to provide further insight in to the geographical variation that exists in the assessment of the patients who are potential candidates for a pelvic exenteration in the hope that it will improve our understanding of these differences and increase the validity of the conclusions that can be drawn from our research on a prospective collaborative basis.

This will be performed by having "real-world" cases selected by our participating centres, anonymising the case and radiological information necessary and by presenting these cases over a series of weeks at MDT meetings all over the world. The data will then be analysed to assess the differences in the ways that certain groups/countries approach the management of these complex and highly varied cases.

ELIGIBILITY:
Inclusion Criteria:

* Complex case from participating PelvEx centre
* Complete clinical information available to allow for informed MDT assessment
* DICOM files for sharing of imaging related to treatment decisions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or recurrent pelvic maligancy who have been treated at a participating PelvEx centre.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Regional/geographic variation in MDT treatment allocations | Through study completion, an average of three months
  Treatment consensus reached for each individual case
Assessment of resectability | Through study completion, an average of three months
  Was the malignancy felt to be resectable by MDT consensus at that institution

SECONDARY OUTCOMES:
Assessment of staging | Through study completion, an average of three months
  Concordance between centres on the TNM staging of disease

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Dublin, Ireland